CLINICAL TRIAL: NCT04533815
Title: Enhancing Sleep Quality for Nursing Home Residents With Dementia: Pragmatic Trial of an Evidence-Based Frontline Huddling Program
Brief Title: Enhancing Sleep Quality for Nursing Home Residents With Dementia
Acronym: 40Winks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Massachusetts, Lowell (Other); The University of Texas Health Science Center, Houston (Other); University of Texas at Austin (Other); Brown University (Other)
Responsible Party: Principal Investigator, A. Lynn Snow, Professor, University of Alabama, Tuscaloosa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R61AG065619-01 (NIH)
Record Dates: First submitted 2020-08-22; First posted 2020-09-01 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease; Dementia; Sleep Disorder; Sleep Disturbance
MeSH Terms: conditions — Alzheimer Disease; Dementia; Sleep Wake Disorders; Parasomnias

STUDY DESIGN:
Intervention Model Description: Pilot study in 3 nursing homes. The pilot phase (R61) informs the next phase (R33), a clinical trial using an incomplete, stepped, wedge cluster randomized controlled trial (RCT) design with 24 nursing homes. Each nursing home in the full clinical trial (R33) will act as its own control (4 staggered steps, with 6 nursing homes per step).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LOCK sleep intervention (Experimental): Nursing home staff receive the LOCK sleep intervention training and thus provide to nursing home residents with dementia the LOCK sleep intervention
  Interventions: Behavioral: LOCK sleep intervention

INTERVENTIONS:
Behavioral: LOCK sleep intervention — Nursing home staff are trained to use a collaborative problem-solving approach to sleep quality improvement using front-line huddling

SUMMARY:
This was a pilot study (R61) to prepare for a full clinical trial (R33) aiming to improve clinical outcomes for an important, growing, and vulnerable population-nursing home (NH) residents with Alzheimer's disease or related dementias (ADRDs). The goal was to pilot and refine the research methods and intervention that would be subsequently evaluated in a full implementation trial (hybrid type III). The goal of the evidence-based intervention (LOCK) that was refined in this pilot study and will be evaluated in the subsequent full clinical trial is to improve the sleep of NH residents with ADRD.

DETAILED DESCRIPTION:
In community (non-VA) NHs [one from each of 3 national NH corporations], the multi-disciplinary research team achieved two aims: (1) refined the LOCK program to focus on sleep for residents with ADRD during this pilot (R61) phase, (2) which prepared the team for the second phase of this two-part NIA-funded grant (the R33 phase) to test the impact and sustainability of this intervention for NH residents with ADRD in an incomplete stepped-wedge randomized controlled trial.

THIS PILOT STUDY R61 PHASE (1 YEAR; N = 3 NHS; 1 NH PER CORPORATION) HAD THE FOLLOWING SPECIFIC AIMS:

1. Refine the LOCK sleep program train-the-trainer protocol by implementing and pilot-testing in three NHs.
2. Test and refine the research methods to: effectively identify eligible NHs and residents; obtain consent; collect primary data from residents and staff (sleep time via actigraph); explore staff impressions of additional sleep measurement devices (Fitbits); transfer primary and secondary data to our data center; and merge all data.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home residents aged >=50 years with an Alzheimer disease or related dementia (ADRD) diagnosis, identified by nursing home staff participating in frontline LOCK sleep huddles as having sleep problems

Exclusion Criteria:

* residents with a high risk of OSA who are not being treated for OSA because actigraph measurements are inaccurate in that population.
* residents who have a persistent bilateral resting tremor or paralysis in both arms (a subset of persons with Parkinson's disease and related significant tremor-causing diagnoses), due to actigraph measurement inaccuracies

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Snow, PhD, Principal Investigator — The University of Alabama
Locations (1):
- The University of Alabama, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share de-identified participant data by depositing data files and associated code books and analysis files with the data repository dataverse (dataverse.org). The research team will follow the University of Alabama IRB guidance and approval for ensuring that the data is appropriately de-identified before posting to dataverse. The IRB-approved informed consent and HIPPAA forms seek participant permission for broad inclusion of participant data for these data sharing and secondary analysis purposes.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within 6 months of study closure, for 5 years
Access Criteria: Under development. Contact PI.

REFERENCES:
- [Background] Snow AL, Loup J, Morgan RO, Richards K, Parmelee PA, Baier RR, McCreedy E, Frank B, Brady C, Fry L, McCullough M, Hartmann CW. Enhancing sleep quality for nursing home residents with dementia: a pragmatic randomized controlled trial of an evidence-based frontline huddling program. BMC Geriatr. 2021 Apr 27;21(1):281. doi: 10.1186/s12877-021-02189-8. PMID 33906631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the three participating community nursing homes. Nursing home staff referred residents to the study that they identified as meeting eligibility criteria.
Period: Overall Study
Arm/Group | LOCK Sleep Intervention
Started | 23
Completed | 16
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Site withdrew | 5

BASELINE CHARACTERISTICS:
Arm/Group | LOCK Sleep Intervention
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.74 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Nighttime sleep minutes (actiwatch measurement) [Mean (Standard Deviation); unit: Nighttime Sleep Minutes] | 520.00 (113.30)

OUTCOME MEASURES:

1. Primary Outcome: Sleep (Actigraph Measurement)
Description: Total sleep time (total minutes asleep each nighttime period - 7pm to 7am)
Time Frame: 15 week sleep intervention period
Population: Enrollees completing the 15-week intervention period
Measure: Mean (Standard Deviation); unit: Nighttime sleep minutes
Arm/Group | LOCK Sleep Intervention
Number analyzed (Participants) | 16
Nighttime sleep minutes | 544.00 (113.97)

ADVERSE EVENTS:
Time Frame: During the active 15-week intervention period for each enrolled resident.
Arm/Group | LOCK Sleep Intervention
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LOCK Sleep Intervention (N=23)
Did not tolerate wearing actiwatch (Social circumstances) | 2 (23) — Participant found watch uncomfortable and communicated desire to have watch removed (either through words or nonverbally by repeatedly pulling at watch)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT04533815/Prot_SAP_000.pdf